CLINICAL TRIAL: NCT06107725
Title: Effect of Oral Minocycline on Acute Stroke Outcome: A Randomized Open Label Prospective Study
Brief Title: Maimonides Minocycline in Stroke Study
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The protocol is in the process to change due to challenges in recruiting participants (without a treatment arm) which is now reflected in 2024-04-01
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Qingliang T. Wang, MD, PhD, Vice Chair of Neurology; Director of Jaffe Comprehensive Stroke Center, Maimonides Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-05-16-MMC
Record Dates: First submitted 2023-10-11; First posted 2023-10-30 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Stroke, Acute; Ischemic Stroke; Hemorrhagic Stroke; Mortality; Morbidity
Keywords: Minocycline; Acute Stroke; Neuroprotection; Mortality; Morbidity; Ischemic stroke; Hemorrhagic Stroke; mRs (Modified Rankin Scale); Clinical outcome
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: Randomized, open label study
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will contact and obtain primary outcome measures of mRS without the knowledge of participants group assignment/treatment received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Stroke Care without Minocycline (No Intervention): 560 Patients will receive standard stroke care.
- Standard Stroke Care with Minocycline (Experimental): 560 patients in the Minocycline arm will receive Minocycline 200 mg every 24 hours for five days with standard stroke care
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Minocycline 200 mg every 24 hours for five days to be initiated within 24hr of stroke onset.
  Arms: Standard Stroke Care with Minocycline

SUMMARY:
The goal of this study is to determine if oral Minocycline's proposed neuroprotective effects further improve the clinical outcomes, including mortality, of acute stroke patients beyond the current standard stroke care in a large scale randomized prospective open label (outcome assessor blinded) clinical trial.

Participants will be randomly assigned (1:1) to take Minocycline 200mg orally every 24 hours for five days, starting within 24 hours from stroke symptoms onset, in addition to standard care or standard care alone.

NIHSS (The National Institutes of Health Stroke Scale) and mRS (Modified Rankin Scale) will be collected at the time of presentation, discharge and again at 30- and 90-days post-discharge. All-cause mortality will also be obtained at 30 days and 90 days.

DETAILED DESCRIPTION:
Studies on animals and humans have shown that Minocycline, a widely used semi-synthetic antibiotic, may protect the brain, spinal cord and nervous system from injuries such as ischemia, trauma, neurodegeneration or inflammation. Minocycline has been shown possibly to reduce the disability and recovery time from stroke.

Hypothesis:

When combined with the standard care treatment, Minocycline's neuroprotective effects improve the clinical outcomes, including the mortality, of acute stroke patients compared to the standard stroke care without Minocycline.

Minocycline 200mg daily, when administered less than 24 hours after onset of acute ischemic stroke orally, improves survival and functional outcome as assessed by improvement of NIHSS - (National Institutes of Health Stroke Scale) score and mRS (Modified Rankin Scale) scores on admission and at discharge (including mortality, mRS=6) and on day 90 post-stroke.

This prospective study will enroll 1120 patients who arrive in the ER at Maimonides Medical Center for suspected acute stroke (excluding transient ischemic attack). After obtaining informed consent, 1120 patients will be enrolled from November 2023 to November 2025. Consecutive randomization will be done, and 560 patients will be assigned to each arm, the Minocycline with Standard care and Standard Care alone arms. The 560 patients in the Minocycline arm will receive Minocycline 200 mg orally every 24 hours for five days in addition to standard care, while the Standard arm will accept only standard care. NIHSS -(National Institutes of Health Stroke Scale) and mRS (Modified Rankin Scale) scores will be collected on presentation, on discharge, and days 30 and 90. A comparison will be made between both arms in both studies for their significance. Statistical analysis will be done with the help of a Maimonides statistician. Interim research will be conducted every six months for outcome significance and safety measures (30-day mortality and symptomatic hemorrhagic conversion).

Subjects:

Patients with clinical suspicion of stroke - both ischemic and hemorrhagic or computer tomography consistent with acute stroke consistent with WHO (World Health Organization) guidelines (excluding transient ischemic attack).

Eligibility Criteria: See below.

Randomization: Consecutive randomization will be done.

Blinding Technique: Outcome assessor-blinded study

Data Collection Procedures:

Patients getting admitted at Maimonides Medical Center from August 2023 for acute stroke will be evaluated, and their eligibility for the trial will be assessed. Then the eligible patients will be randomly assigned to the Minocycline or the Standard group in their respective arms consecutively. Acute Ischemic and Hemorrhagic patients will be treated with Minocycline along with standard care versus standard care alone. Patient demographic details and information on co-morbidities are collected. Their NIHSS (National Institutes of Health Stroke Scale) and mRS (Modified Rankin Scale) scores will be measured at the time of presentation and discharge and again at 30- and 90-days post-discharge. All-cause mortality will also be obtained at 30 days and 90 days. The outcomes are documented, and the results will be analyzed.

Data Analysis:

Data analysis will be performed with the assistance of the Maimonides Medical Center biostatistician. All numeric variables will be summarized with mean and 95% confidence interval where appropriate and median and IQR (Interquartile range) (if necessary. All categorical variables will be summarized with frequency and percentage. Continuous variables that are risk factors or demographics will be compared across groups using a t-test or Wilcoxon rank sum test. Categorical risk factors and demographics will be compared between groups using a chi-square or fisher exact test.

The primary outcome of reduced NIHSS (National Institutes of Health Stroke Scale) and mRS (Modified Rankin Scale) as discharge will be evaluated using a student's T-test (to compare the means between two groups). The outcome of mortality will be evaluated using a Fisher exact test. 90-day outcomes will be evaluated similarly. To control for additional risk factors, including baseline NIHSS (National Institutes of Health Stroke Scale) and mRS (Modified Rankin Scale), the study team will also create a generalized linear model with a normal link function for continuous outcomes, controlling for risk factors significantly different between groups. For mortality, the investigators will use a generalized liner model with a logistic link function to control for risk factors that varied considerably between groups.

Target power : 0.8 Actual power : 0.800 Alpha : 0.05 Assumed population means : 3.2 for the placebo group and 2.9 for the Minocycline group (with an expected difference between the population's means is 0.51) Calculated size : 560 in each arm with a total of 1120 patients after considering a 10% attrition rate.

Expected Outcomes:

When combined with the standard care treatment, Minocycline's neuroprotective effects improve the clinical outcomes, including the mortality, of acute stroke patients compared to routine stroke care without Minocycline.

Time Period:

Once IRB approval is obtained, the investigator expects to start subject enrollment on November 1st, 2023, followed by chart review, data collection, and analysis to begin and be completed within 27 months on Feb 1st, 2026 (including 3 months for outcome measures collection and data analysis after last enrolled patient). The investigator aims to achieve the above process in an expedited manner, as the results will be used for performance improvement and publications. Interim analyses including safety monitoring will be conducted at 25%, 50%, and 75% enrollment intervals by the study team and an independent DSMB (Data and Safety Monitoring Board).

ELIGIBILITY:
Inclusion Criteria:

1. Age >/=18
2. Acute onset neurological deficit consistent with acute ischemic stroke or on imaging consistent with acute ischemia as defined by WHO (World Health Organization) guidelines
3. Acute onset of neurological deficits with intracerebral Hemorrhage on imaging consistent with intracerebral bleed
4. The onset of symptoms less than 24 hours
5. Measurable neurological deficit using NIHSS (National Institutes of Health Stroke Scale )

Exclusion Criteria:

1. Clinically not suspect stroke.
2. Allergic to the Tetracycline group of medications or Intolerance to Minocycline
3. Pregnancy or suspected pregnancy
4. Previous history of intolerance to minocycline
5. Acute or chronic renal failure
6. Any patients with contraindications to undergo CT/ MRI
7. Life expectancy less than one year or severe co-morbidities or comfort measure only (CMO) on admission
8. Pre-existing infectious disease requiring antibiotics
9. Inability to tolerate enteral medications/feeds
10. Patient/ family refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Stroke Care Without Minocycline | Standard Stroke Care With Minocycline
Started | 0 | 2
Completed | 0 | 0
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: The study was terminated after 2 patients were enrolled in the study. No patients were enrolled in the without Minocycline group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Stroke Care Without Minocycline | Standard Stroke Care With Minocycline | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 2 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: In-hospital and 30-day Mortality
Description: Mortality rates during hospitalization and at 30 days
Time Frame: 30 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Stroke Care Without Minocycline | Standard Stroke Care With Minocycline
Number analyzed (Participants) | 0 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: The study was terminated after 2 patients were enrolled in the study. No patients were enrolled in the without Minocycline group.
Arm/Group | Standard Stroke Care Without Minocycline | Standard Stroke Care With Minocycline
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT06107725/Prot_SAP_000.pdf